CLINICAL TRIAL: NCT07231055
Title: Virtually Designed Custom-Made Titanium Plate Versus Three-Dimensional Lambda Plate for Management of Mandibular Subcondylar Fractures: (A Randomized Controlled Trial)
Brief Title: Comparative Trial of Custom-Made Titanium Plates Versus 3D Lambda Plates for Mandibular Subcondylar Fractures
Acronym: SUBCONDPLATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Ahmed Thamer Al Masoud, Sponsor-Investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TU-OMFS-2025-SUBCONDYLAR-CT
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Mandibular Sub-condylar Fracture
Keywords: Mandibular sub-condylar fractures; Fractures of mandible; condylar fractures of mandible; Patient specific plate; CAD/CAM; Virtual Surgical planning; Randomized Controlled trial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Custom-Made plate Group (Experimental): Patient-specific titanium plate fabricated using virtual surgical planning, CT-based segmentation, and 3D design for fixation of mandibular subcondylar fractures.
  Interventions: Device: Custom-Made Plate Group
- Three-Dimensional (3D) Lambda plate Group (Active Comparator): Standard ready-made three-dimensional titanium lambda plate used for open reduction and internal fixation of mandibular subcondylar fractures.
  Interventions: Device: Three-Dimensional Lambda Plate

INTERVENTIONS:
Device: Custom-Made Plate Group — Virtually designed Patient-specific titanium plate fabricated using virtual surgical planning, CT-based segmentation, and 3D design for fixation of mandibular subcondylar fractures.
  Arms: Custom-Made plate Group
Device: Three-Dimensional Lambda Plate — Standard ready-made three-dimensional titanium lambda plate used for open reduction and internal fixation of mandibular subcondylar fractures.
  Arms: Three-Dimensional (3D) Lambda plate Group

SUMMARY:
This randomized clinical trial compares virtually designed custom-made titanium plates with conventional three-dimensional (3D) lambda plates for the fixation of mandibular subcondylar fractures. A total of 24 fracture sites will be treated using a retromandibular trans-masseteric approach and evaluated through virtual surgical planning, radiographic analysis, and functional outcomes. The study aims to determine whether customized plates provide superior anatomical accuracy, stability, and recovery compared with standard 3D plates.

DETAILED DESCRIPTION:
Mandibular subcondylar fractures can affect occlusion, mandibular function, and facial symmetry, and remain a topic of ongoing clinical debate regarding optimal fixation methods. Conventional management often relies on standardized three-dimensional (3D) plates, such as the lambda configuration, which provides reliable fixation but may not precisely conform to the individual patient's anatomy.

Advances in virtual surgical planning (VSP) and computer-aided design now allow for the fabrication of patient-specific titanium plates that follow the exact contours of each patient's mandibular anatomy. These customized implants may improve reduction accuracy, minimize inter-fragmentary gaps, enhance postoperative stability, and reduce intraoperative manipulation.

In this study, 24 subcondylar fracture sites will be randomly assigned to either a patient-specific custom-made plate group or a conventional 3D lambda plate group. All procedures will be performed using the retromandibular trans-masseteric approach. Preoperative planning will include CT-based segmentation, virtual fracture reduction, and 3D model generation. Postoperative follow-up will be conducted at multiple intervals to assess radiographic bone healing, condylar and gonial width symmetry, inter-fragmentary gap, mandibular function, pain scores, occlusion, edema, and soft tissue healing.

The study seeks to evaluate whether the use of a customized fixation system results in measurable improvements in surgical precision and functional recovery compared with standard 3D plating techniques. Findings from this clinical trial may support evidence-based decision-making in the selection of fixation systems for subcondylar fractures and clarify the potential clinical benefits of patient-specific implant technology.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients with mandibular subcondylar fracture indicated for open reduction and internal fixation.

Exclusion Criteria:

* Patients with systemic diseases that affect tissue healing.
* Mandibular condylar head or neck fractures. (Condylar neck is the where the caudal portion of the joint capsule attaches. It is the thin constricted area immediately below the condylar head.)

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-12-28 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-10-29 (Actual)

PRIMARY OUTCOMES:
Operative time | Intraoperative (recorded during the surgical procedure)
  The total operative time required to perform open reduction and internal fixation of mandibular subcondylar fractures, measured from incision to completion of fixation. The outcome will be compared between the custom-made titanium plate group and the 3D lambda plate group.

SECONDARY OUTCOMES:
Pain Scor (VAS) | Immediate postoperative, 1 week, 2 weeks, 1 month, 3 months, 6 months.
  Visual Analog Scale score to assess postoperative pain intensity over time.
Occlusal Function (Uglesic Score) | 1 week, 1 month, 3 months, 6 months.
  Evaluation of occlusal stability and masticatory function using the Uglesic et al. (1993) occlusion questionnaire.
Mouth Opening (Maximum Inter-Incisal Distance, mm) | Preoperative, 1 week, 2 weeks, 1 month, 3 months, 6 months.
  Measurement of maximal mouth opening to evaluate functional recovery.
Radiographic Bone Healing (Computed Tomography Evaluation) | 1 month, 3 months, 6 months.
  Computed Tomography based evaluation of bone union, accuracy of reduction and consolidation at the fracture site.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A Almasoud, Principal Investigator — Faculty of Dentistry, Tanta University, Egypt; Mohamed M Khedr, Principal Investigator — Faculty of Dentistry, Tanta University, Egypt; Ahmed A Mosleh, Principal Investigator — Faculty of Dentistry, Tanta University, Egypt
Locations (1):
- Faculty of Dentistry, Tanta University., Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No